CLINICAL TRIAL: NCT06379087
Title: Prospective Phase II Study of Hypofractionated Radiotherapy Sequential Tislelizumab and Anlotinib in the Neoadjuvant and Adjuvant Therapy for Stage II-IIIA Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy Followed by Tislelizumab and Anlotinib Aeoadjuvant/Adjuvant Therapy for Stage II-IIIA NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ji Yongling (Other)
Responsible Party: Sponsor-Investigator, Ji Yongling, Physician, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-PIONEER
Record Dates: First submitted 2024-04-11; First posted 2024-04-23 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; tislelizumab; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Neoadjuvant therapy regimen (2 cycles):
  1. Receive 3-day hypofractionated treatment on Day 1, Day 2, and Day 3, with a total dose of 24Gy (8Gy*3).
  2. Within 1 week after radiotherapy, receive neoadjuvant tislelizumab (200 mg, intravenous drip, d1) combined with anlotinib (10 mg, oral, D1-14) . Each 3 weeks is a medication cycle.
  Surgical protocol: The surgical approach was determined by the surgeon according to the patient's condition, including but not limited to thoracoscopic/open lobectomy/sleeve lobectomy/combined lobectomy/pneumonectomy. Lymph node dissection requires at least three stations of mediastinal lymph node dissection.
  Adjuvant therapy regimen: tislelizumab (200 mg, intravenous drip, d1) combined with Anlotinib (10 mg, oral, D1-14). Each 3 weeks is a medication cycle, for 1 year.
  Interventions: Drug: Anlotinib Hydrochloride Capsule; Drug: Tislelizumab Injection; Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor that inhibits both tumor angiogenesis and tumor cell proliferation by blocking VEGFR, FGFR, PDGFR, and c-Kit simultaneously.
  Other Names: Anlotinib
Drug: Tislelizumab Injection — Tislelizumab is a humanized IgG4 anti-PD-1 monoclonal antibody.
  Other Names: Tislelizumab
Radiation: Hypofractionated Radiotherapy — Hypofractionated Radiotherapy Extent of radiotherapy: Primary lesion in the lung. Radiotherapy technique: IGRT. Radiotherapy delivery equipment: linear accelerator or TOMO accelerator or CyberKnife.

SUMMARY:
This study is a single-center, prospective, single-arm exploratory clinical study of hypofractionated radiotherapy followed by tislelizumab and anlotinib neoadjuvant and adjuvant therapy. It is designed for patients with stage II-IIIA non-small cell lung cancer. The efficacy and safety of hypofractionated radiotherapy sequential tislelizumab and anlotinib in the neoadjuvant and adjuvant treatment of stage II-IIIA non-small cell lung cancer are observed. Finally, it provides new evidence-based medical evidence for the perioperative treatment of non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is a single-center, prospective, single-arm, exploratory clinical study aimed at evaluating the efficacy and safety of hypofractionated radiotherapy sequential tislelizumab and anlotinib in the neoadjuvant and adjuvant treatment of stage II-IIIA non-small cell lung cancer. If the subject does not voluntarily withdraw from the trial, or the toxic and side effects caused by the drug are intolerable, or the investigator considers that the subjects are not suitable for further trials, each subject will receive the following treatments before and after surgery, and the efficacy evaluation and follow-up will be performed in each cycle.

After completing all screening activities, eligible patients will enter the study and receive the following treatment and visits: First, receive 24 Gy (8 Gy*3) of hypofractionated treatment on d1-3 after the start of the study, and then receive neoadjuvant therapy with tislelizumab combined with anlotinib within 1 week after radiotherapy. Each 3 weeks is a medication cycle, for a total of 2 cycles. Patients will undergo radical surgery after neoadjuvant treatment, and then receive tislelizumab and anlotinib adjuvant treatment after surgery. Each 3 weeks is a medication cycle, and it is maintained for 1 year. The 1-year event-free survival (EFS) rate, complete pathological response (pCR) and major pathological response (MPR) were evaluated to evaluate the safety of medical/surgical treatment for patients.

Neoadjuvant therapy regimen (2 cycles):

1. Receive 3-day hypofractionated treatment on Day 1, Day 2, and Day 3, with a total dose of 24Gy (8Gy*3).
2. Within 1 week after radiotherapy, receive neoadjuvant tislelizumab (200 mg, intravenous drip, d1) combined with anlotinib (10 mg, oral, D1-14) . Each 3 weeks is a medication cycle.

Surgical protocol: The surgical approach was determined by the surgeon according to the patient's condition, including but not limited to thoracoscopic/open lobectomy/sleeve lobectomy/combined lobectomy/pneumonectomy. Lymph node dissection requires at least three stations of mediastinal lymph node dissection.

Adjuvant therapy regimen: tislelizumab (200 mg, intravenous drip, d1) combined with Anlotinib (10 mg, oral, D1-14). Each 3 weeks is a medication cycle, for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 18-75 years old;
* (2) Early stage II-IIIA NSCLC (AJCC 8th edition), NSCLC, confirmed in tissue (AJCC eighth edition);
* (3) All lesions are assessed to be eligible for surgical resection;
* (4) The primary tumor can be treated with hypofractionated radiotherapy after evaluation;
* (5) Epidermal growth factor receptor/anaplastic lymphoma kinase/ROS1 gene fusions mutation was negative in primary tumor or lymph node metastasis;
* (6) ECOG PS score: 0~1;
* (7) Expected survival more than 1 year;
* (8) At least one measurable lesion (RECIST 1.1);
* (9) Females of childbearing potential should agree to use contraceptive measures (such as intrauterine device, contraceptives or condoms) during the study and within 3 months after the end of the study; have a negative serum or urine pregnancy test within 7 days before study enrollment and must be non-lactating subjects; and males should agree to use contraceptive measures during the study and within 3 months after the end of the study period;
* (10) Subjects voluntarily participate in this study, sign the informed consent form and had good compliance;
* (11) Subjects are suitable after MDT discussion.

Exclusion Criteria:

Participants with any of the following criteria were excluded from the trial:

* (1) The location of the primary tumor was assessed by the radiologist and considered unsuitable for hypofractionated therapy;
* (2) The pathological type is small cell lung cancer, or mixed tumor with small cell components;
* (3) A history of or concurrent with other malignancies;
* (4) Received any anti-tumor treatment before this study, including chemotherapy, radiotherapy, targeted therapy (including but not limited to monoclonal antibodies, small molecule tyrosine kinase inhibitors, etc.) and immunotherapy;
* (5) The Imaging (CT/MR/PET-CT) showed tumor invasion of great vessels or blurred boundary with blood vessels, or the presence of any pulmonary cavity or necrotic lesions;
* (6) Hemoptysis, active bleeding, ulcer, intestinal perforation, intestinal obstruction within 3 months before enrollment;
* (7) Previous interstitial lung disease, drug-induced interstitial disease or any clinical evidence of active interstitial lung disease; baseline CT scan found idiopathic pulmonary fibrosis;
* (8) According to the investigator's judgment, there are serious or uncontrollable systemic diseases (such as unstable or uncompensated respiratory, cardiac, hepatic or renal diseases) or any unstable systemic diseases (including active infection, grade III hypertension, unstable angina, congestive heart failure, liver and kidney or metabolic diseases);
* (9) Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs acting on another co-inhibitory T cell receptor (e.g., CTLA-4, OX-40, CD137);
* (10) The presence of uncontrollable third space effusion, such as a large number of pleural effusion or ascites or pericardial effusion;
* (11) Urine routine showed urine protein ≥ + +, or 24h urine protein ≥ 1g or severe liver and kidney dysfunction;
* (12) Uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
* (13) Subjects requiring systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive agents within 14 days before the first dose;
* (14) Hyperactive/venous thrombotic events occurred within 6 months, such as cerebrovascular accident (including cerebral hemorrhage, cerebral infarction, temporary ischemic attack, etc.);
* (15) Excessive surgery or significant trauma within 28 days before enrollment;
* (16) Pregnant or lactating women;
* (17) Subjects who are considered to be unsuitable for enrollment for other reasons according to the judgment of the investigators..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR Rate | 12 months
  Complete pathological response (pCR), defined as the proportion of patients in the ITT analysis set and surgical population analysis set who have no residual tumor in the resected primary tumor and metastatic lymph nodes as assessed by the investigator after the completion of neoadjuvant therapy. Patients who do not meet these criteria, including those who do not undergo surgical resection, will be considered non-responders.

SECONDARY OUTCOMES:
1-year EFS Rate | Baseline up to 1 years
  1-year EFS rate is defined as the proportion of patients who have not experienced radiographic disease progression, local recurrence or distant metastasis, or death due to any cause assessed by the investigator according to RECIST 1.1 Version, from enrollment to 1 year in the intent-to-treat (ITT) analysis set. The 1-year EFS rate is evaluated by the Kaplan-Meier (KM) method.
MPR Rate | 12 months
  Major pathological response (MPR) was defined as the proportion of patients in the ITT analysis set and surgical population analysis set with ≤ 10% residual viable tumor cells in the resected primary tumor and metastatic lymph nodes after the completion of neoadjuvant therapy as assessed by the investigator. Patients who do not undergo surgical resection for reasons such as disease progression will be considered non-responders.
Adverse Events (AEs) according to CTCAE (V5.0) (Safety Evaluation) | Baseline up to 3 years
  The number of abnormal data on potential adverse reaction

CONTACTS AND LOCATIONS:
Overall Officials: YongLing Ji, PhD, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No